CLINICAL TRIAL: NCT00330980
Title: Statins and Noncardiovascular Endpoints
Brief Title: Effects of Statin Medications on Mental Processes, Behavior, and Serotonin Levels
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Beatrice A. Golomb, MD, PhD, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 394; R01HL063055 (NIH)
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2008-07

CONDITIONS: Dyslipidemias
Keywords: Cognition; Statins; Serotonin; Cholesterol
MeSH Terms: conditions — Dyslipidemias | interventions — Pravastatin; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental): Participants will receive 20 mg of simvastatin for 6 months.
  Interventions: Drug: 20 mg Simvastatin
- 2 (Experimental): Participants will receive 40 mg of pravastatin for 6 months.
  Interventions: Drug: 40 mg Pravastatin (Pravachol)
- 3 (Placebo Comparator): Participants will receive placebo for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 40 mg Pravastatin (Pravachol) — Participants will receive 40 mg of pravastatin for 6 months.
  Arms: 2
Drug: 20 mg Simvastatin — Participants will receive 20 mg of simvastatin for 6 months.
  Arms: 1
Drug: Placebo — Participants will receive placebo for 6 months.
  Arms: 3

SUMMARY:
Statins are cholesterol-lowering medications that are often prescribed for individuals with high cholesterol and who are at risk for heart disease. Preliminary research has shown that statins may have other effects on the body that are unrelated to the heart. The purpose of this study is to evaluate the impact of statins on mood, mental processes, aggression, and serotonin levels.

DETAILED DESCRIPTION:
Individuals at risk for coronary artery disease are often prescribed statins, which are medications that reduce the amount of cholesterol in the blood. By lowering cholesterol levels, these individuals have a lower incidence of heart disease, heart attacks, and stroke. Simvastatin and pravastatin are two common statins that are often prescribed for individuals with high cholesterol. While statins are effective at lowering cholesterol levels, their effect on mood, behavior, and aggression has not been widely studied. Preliminary research has shown that lowering cholesterol levels may lead to an increase in aggressive behaviors and a change in cognitive function. Serotonin, a type of neurotransmitter, is believed to play an important role in the regulation of mood, as well as behavior and cognition. The direct effect of statins on serotonin levels remains unknown. The purpose of this study is to evaluate the effect of simvastatin and pravastatin on mood, cognition, aggression, and serotonin levels.

This study will enroll individuals who do not currently take cholesterol-lowering medications. Participants will be randomly assigned to receive 20 mg of simvastatin, 40 mg of pravastatin, or placebo for 6 months. Study visits will occur at baseline and Months 1, 3, 6, and 8. Height, weight, and waist circumference will be measured at all study visits. Blood and urine will be collected for laboratory testing, and standardized psychological questionnaires will assess cognition, aggression, mental flexibility, memory, depression, sleep quality, and quality of life at Months 1, 6, and 8. At Month 3, medication side effects will be monitored and a liver function test will be performed. Participants' partners will take part in a telephone interview at this time. At baseline and Month 6, some participants will undergo cardiac reactivity testing. During this procedure, participants will be videotaped and monitored for vital sign changes (blood pressure and heart rate) while they talk about potentially stressful situations.

ELIGIBILITY:
Inclusion Criteria:

* LDL cholesterol level between 115-190 mg/dL
* Able to fast prior to blood draw
* Able to comfortably read and write in English
* Able and willing to refrain from donating whole blood during study participation
* Willing to abstain from consuming large amounts of grapefruit juice

Exclusion Criteria:

* Current use of lipid-lowering medications
* Symptomatic atherosclerotic disease, such as coronary artery disease, kidney failure or insufficiency, peripheral arterial disease, or cerebrovascular disease
* Cancer
* HIV infected
* Medical or psychiatric condition that prevents full study participation or follow-up (e.g., active psychosis)
* Active liver disease or unexplained persistent elevated transaminase levels
* Major surgery or hospitalization in the 3 months prior to study entry
* Current use of cyclosporin, erythromycin, clarithromycin, nefazodone, or any "azole" antifungals, including fluconazole, itraconazole, ketoconazole, mibefradil, or protease inhibitors
* Female of childbearing potential
* Current participation in another clinical trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2000-04; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Effects of statins on cognition, serotonin biochemistry, and aggression | Measured at Months 6 and 8

SECONDARY OUTCOMES:
Effect of statins on mood, and other cognitive, behavioral, and biochemical measures | Measured at Months 6 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice A. Golomb, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

REFERENCES:
- [Background] Golomb BA, Criqui MH, White HL, Dimsdale JE. The UCSD Statin Study: a randomized controlled trial assessing the impact of statins on selected noncardiac outcomes. Control Clin Trials. 2004 Apr;25(2):178-202. doi: 10.1016/j.cct.2003.08.014. PMID 15020036
- [Background] Golomb BA, Criqui MH, White H, Dimsdale JE. Conceptual foundations of the UCSD Statin Study: a randomized controlled trial assessing the impact of statins on cognition, behavior, and biochemistry. Arch Intern Med. 2004 Jan 26;164(2):153-62. doi: 10.1001/archinte.164.2.153. PMID 14744838
- [Derived] Golomb BA, Dimsdale JE, Koslik HJ, Evans MA, Lu X, Rossi S, Mills PJ, White HL, Criqui MH. Statin Effects on Aggression: Results from the UCSD Statin Study, a Randomized Control Trial. PLoS One. 2015 Jul 1;10(7):e0124451. doi: 10.1371/journal.pone.0124451. eCollection 2015. PMID 26132393
- [Derived] Golomb BA, Chan VT, Evans MA, Koperski S, White HL, Criqui MH. The older the better: are elderly study participants more non-representative? A cross-sectional analysis of clinical trial and observational study samples. BMJ Open. 2012 Dec 14;2(6):e000833. doi: 10.1136/bmjopen-2012-000833. Print 2012. PMID 23242479
- [Derived] Golomb BA, Koperski S, White HL. Association between more frequent chocolate consumption and lower body mass index. Arch Intern Med. 2012 Mar 26;172(6):519-21. doi: 10.1001/archinternmed.2011.2100. No abstract available. PMID 22450943
- [Derived] Golomb BA, Evans MA, White HL, Dimsdale JE. Trans fat consumption and aggression. PLoS One. 2012;7(3):e32175. doi: 10.1371/journal.pone.0032175. Epub 2012 Mar 5. PMID 22403632
- [Derived] Golomb BA, Dimsdale JE, White HL, Ritchie JB, Criqui MH. Reduction in blood pressure with statins: results from the UCSD Statin Study, a randomized trial. Arch Intern Med. 2008 Apr 14;168(7):721-7. doi: 10.1001/archinte.168.7.721. PMID 18413554